CLINICAL TRIAL: NCT02217202
Title: Prospective Cohort Study of the AQUACEL™ Ag SURGICAL Cover Dressing in Total Knee Replacement Surgery
Brief Title: Study of AQUACEL™ Ag Surgical Cover Dressing Following Total Knee Replacement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn before ethical approval granted
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Alistair Ewen, Orthopaedic Researcher, Golden Jubilee National Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ortho 1302
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis
Keywords: knee replacement; knee arthroplasty; revision; high risk
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ConvaTec Ag (Experimental): Use of ConvaTec Ag sugical cover dressing post-operatively until wound has healed.
  Interventions: Device: Aquacel Ag dressing

INTERVENTIONS:
Device: Aquacel Ag dressing — Participants will have their knee arthroplasty wound dressed using the Aquacel Ag dressing instead of the standard Aquacel dressing.
  Other Names: Convatec Aquacel Ag dressing

SUMMARY:
The aim of the study is to determine whether the AQUACEL™ Ag SURGICAL cover dressing is successful in reducing the incidence of wound infection in high risk patients following total knee replacement. We will also look at the status of the wound, occurrence of blistering, biochemistry results, dressing wear time and the number of dressing changes to quantify the dressing performance.

DETAILED DESCRIPTION:
All eligible patients over a two month period will be identified and invited to take part in the study. Identification will be done though examination of clinical case notes of patients who are candidates for total knee replacement or revision surgery. Demographic and medical history data for all study patients will be collected. This will include age, gender, BMI, smoking habits, alcohol consumption, diagnosis, operation, laterality and comorbidities. All eligible patients who fulfil the selection criteria will be informed of the study at their pre-surgery consultation, provided with the patient information sheet and approached to take part in the study at a later date.

Patients who have agreed to take part in the study will have their knee surgery performed in the same manner as if they had not agreed to take part. The clinical team will be informed of a patient's participation in the study and will ensure that the AQUACEL™ Ag SURGICAL cover dressing is used instead of the standard dressing protocol with these patients, both immediately after surgery and at any other time when the patient requires the dressing to be changed before discharge. Study patients will also be given a sufficient supply of the dressing for home use on discharge from the hospital.

Patients will be observed during their inpatient stay where data including the wound status, occurrence of blistering, dressing wear time, number of dressing changes, ease of dressing changes, any unforeseen side effects and any surgical site infection will be recorded to quantify the dressing performance by the healthcare staff. Appropriate data from lab results will be extracted. After discharge, data will be collected from the Prevention and Control of Infection team at regular intervals up to 30 days postoperatively. Study patients will be followed up, as per hospital protocol, at six weeks by the Arthroplasty Outcomes team. Data from this follow up will also be included in the study. After this appointment, patients will no longer have any involvement in the study.

Once the data set is completed statistical analysis will be carried out to compare the results of this study with those of a retrospective cohort study of a similar patient group, where the Jubilee method dressing (a combination of DuoDERM® and AQUACEL® was used).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40
* Revision of total knee replacement
* Rheumatoid arthritis or secondary arthritis
* Patients on Warfarin
* Patients on steroids
* Patients on long term antibiotics
* Previous deep joint infection

Exclusion Criteria:

* Allergy to silver
* Simultaneous bilateral total knee replacement patients
* Patients who do not wish to participate
* Patients who are unable to give informed consent
* Patients who are unable to attend Golden Jubilee National Hospital for follow up

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2050-01 (Estimated); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infections. | Up to 6 weeks post-operatively.
  What is the incidence of surgical site infections following total knee replacements and revisions in high risk patients when using the AQUACEL™ Ag SURGICAL cover dressing?

SECONDARY OUTCOMES:
Dressing performance. | Up to 6 weeks post-operatively.
  How does the AQUACEL™ Ag SURGICAL cover dressing perform in terms of the occurrence of blistering, dressing wear time and the number of dressing changes, ease of use and number of unforeseen complications?

CONTACTS AND LOCATIONS:
Overall Officials: Alistair M Ewen, PhD, Principal Investigator — Golden Jubilee National Hospital